CLINICAL TRIAL: NCT06483295
Title: Randomized Controlled Study on Improving Patient-reported Outcomes After Lung Cancer Surgery With Mobile Internet Platform
Brief Title: Improving Patient-reported Outcomes After Lung Cancer Surgery With Mobile Internet Platform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xinghua Cheng, Director, Head of Oncology Surgery, Clinical Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ShanghaiChestPRO
Record Dates: First submitted 2024-03-13; First posted 2024-07-03 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: patient-reported outcomes; Internet
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Mobile Internet Platform Follow-up Group
  Interventions: Other: Using mobile internet platforms for follow-up management of postoperative symptoms in lung cancer patients.
- Group B (No Intervention): Traditional Outpatient Follow-up Group

INTERVENTIONS:
Other: Using mobile internet platforms for follow-up management of postoperative symptoms in lung cancer patients. — Using mobile internet platforms for follow-up management of postoperative symptoms in lung cancer patients.
  Arms: Group A

SUMMARY:
This study focuses on the significant impact of lung cancer in China, highlighted by its high incidence and mortality rates, influenced by factors like aging populations, smoking, and environmental issues. It emphasizes the importance of understanding the duration, severity, and factors affecting post-surgery symptoms like pain and coughing in patients. The research underlines the value of patient-reported outcomes (PROs) in enhancing postoperative care and survival rates through improved symptom monitoring and patient engagement. Utilizing internet technology, specifically a platform integrated with WeChat, the study aims to improve patient management and follow-ups post-discharge. The objective is to use mobile internet technology to build a high-quality prospective database on postoperative lung cancer patient outcomes, analyzing factors affecting postoperative discomfort and assessing the role of interactive platforms in improving patient care.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related deaths worldwide. In China, it has become the malignancy with the highest incidence and mortality rates, exacerbated by aging populations, smoking, and environmental issues. Post-major lung surgery, patients often experience reduced quality of life due to symptoms like pain and coughing. However, the duration, severity, and factors influencing these symptoms during recovery are not fully understood. Notably, recent attention has been given to the direct collection of patient-reported outcomes (PROs) for subjective symptom monitoring and improving patient care. Incorporating PRO monitoring in cancer patient follow-ups can reduce postoperative discomfort, enhance treatment tolerance and adherence, detect early relapses, and improve survival rates. Internet technology significantly expands information exchange frequency and efficiency. Management platforms based on internet mobile applications can enhance patient management compliance, enable intelligent follow-ups, and strengthen doctor-patient interaction. The investigators' hospital intends to utilize its internet hospital platform, integrated with WeChat (a Tencent application in China), for assisting in-patient management and post-discharge surveillance through automated multimedia material and PROs. WeChat, similar to Facebook and WhatsApp, is a multifunctional messenger app with over a billion active monthly users in China, effectively using an application already familiar to patients rather than introducing new ones.

This study aims to leverage mobile internet technology to transform traditional database construction, enhance the efficiency and accuracy of prospective database information collection, and establish a high-quality prospective database of postoperative lung cancer patient-reported outcomes. This will facilitate the analysis of factors influencing postoperative discomfort in patients and explore the role of interactive mobile internet technology platforms in improving postoperative PROs, thereby elevating the diagnostic and treatment standards in this field.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Stage I-III lung cancer and surgically resected at our centre.
2. Owns and uses a smartphone and can use WeChat.
3. Volunteer to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Received any non-surgical anti-tumour therapy (radiotherapy, chemotherapy, targeted therapy or immunotherapy) for lung cancer during the follow-up period.
2. After enrolment, preoperative emergence of serious comorbidities (inability to tolerate surgery or anaesthesia) that are not suitable for, or cannot be implemented as planned, in the study's treatment regimen.
3. After admission, the patient's condition changes and the need to change from elective surgery to emergency surgery is confirmed by the doctor in charge.
4. At any stage after entering the study, the patient voluntarily requests to withdraw or discontinue treatment due to personal reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
complaints of discomfort | 4 months
  MDASI-LC score for complaints of discomfort at postoperative months 1, 3 and 4
  Postoperative discomfort chief complaint MDASI-LC score:
  Choose a number from 0 (asymptomatic) to 10 (the most severe level imaginable) for each item to indicate the severity of the symptoms.
  The main complaints of postoperative discomfort include: pain, cough, shortness of breath (key points) Other factors include fatigue, nausea, insomnia, depression, memory loss, loss of appetite, drowsiness, dry mouth, sadness, vomiting, numbness or stinging wounds, constipation, etc

SECONDARY OUTCOMES:
Life quality | 4 months
  Quality of life scores at postoperative months 1, 3, and 4
  EQ5D scoring table for postoperative quality of life:
  Q1: Activity ability A: Walking is not a problem; B: There are some walking problems; C: Bedridden and unable to get up.
  Q2: Self care ability A: Can be completely self-care; B: There are some issues with taking a shower or dressing; C: Unable to take a shower or dress on their own.
  Q3: Daily activities (such as work, study, household chores, family or leisure activities) A: There is no problem with daily activities; B: There are some issues with daily activities; C: Unable to perform daily activities Q4: Pain/discomfort A: No pain/discomfort; B: Moderate pain/discomfort; C: Extreme pain/discomfort Q5: Anxiety/Depression A: Not anxious/depressed; B: Mild anxiety/depression; C: Moderate anxiety/depression
Pulmonary function-the absolute value of FEV1 | 4 months
  Pulmonary function test results comparing different resection styles
  Perform lung function tests during the study period, including the absolute value of FEV1, the percentage of FEV1 to expected values, etc
Pulmonary function-the percentage of FEV1 to expected values | 4 months
  Pulmonary function test results comparing different resection styles
  Perform lung function tests during the study period, including the absolute value of FEV1, the percentage of FEV1 to expected values, etc
Change of breath sounds | 4 months
  Modelling of breath sounds after resection of different resection styles
  By collecting postoperative respiratory sounds from different resection methods, converting the audio into digital signals for analysis, and then modeling and calculating, a large model of postoperative respiratory sounds from different resection methods is established to evaluate the postoperative respiratory sounds of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Cheng, MD, Principal Investigator — Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China.
Locations (1):
- Zuodong Song, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Luo Y, Cheng Y, Song Z, Chen H, Bo Y, Shixing H. Patient-reported outcomes with a personalized follow-up program after lung cancer resection: A single-center randomized controlled trial. Asia Pac J Oncol Nurs. 2026 Jan 2;13:100844. doi: 10.1016/j.apjon.2025.100844. eCollection 2026 Dec. PMID 41625083